CLINICAL TRIAL: NCT04684875
Title: A Prospective, Multi-center, Non-Randomized Study to Evaluate the Quality of Life Impact and Symptoms After Treatment Using Low Power Radiofrequency Energy Applied to the Posterior Nasal Nerve Area for Symptomatic Relief of Chronic Rhinitis
Brief Title: Quality of Life Impact of Chronic Rhinitis Treatment With Aerin Medical Device
Status: Completed | Type: Observational
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CTP1078
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Chronic Rhinitis
Keywords: Chronic rhinitis; Posterior nasal nerve; Quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Long-Term Study Subjects: All subjects who were treated with the Aerin Medical InSeca/RhinAer Stylus in the 50-subject TP668 interventional study, who consent to continue to provide quality of life data.
  Interventions: Device: Radiofrequency Stylus

INTERVENTIONS:
Device: Radiofrequency Stylus — Low power radiofrequency energy delivered to the posterior nasal nerve area
  Other Names: Aerin Medical Device; InSeca Stylus; RhinAer Stylus

SUMMARY:
Evaluation of long-term (2-year) quality of life and symptoms after chronic rhinitis treatment with the Aerin InSeca/RhinAer Stylus

DETAILED DESCRIPTION:
This is a prospective, non-randomized, multicenter follow-up study to collect long-term data on a cohort of patients who participated in the Aerin Medical TP668 study, "Clinical Evaluation of Low Power Radiofrequency Energy Applied to the Posterior Nasal Nerve Area for Symptomatic Relief of Chronic Rhinitis". The study will be conducted in a maximum of 5 centers that participated and enrolled patients in the TP668 study.

ELIGIBILITY:
Inclusion Criteria:

* Received treatment for chronic rhinitis in Aerin Study TP668

Exclusion Criteria:

* Unwilling to participate in this long-term study

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who completed the 52-week follow-up visit of Aerin Study TP668 and consent to provide long-term quality of life and symptom information.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline rTNSS | 24 months
  Mean change in reflective Total Nasal Symptom Score (rTNSS) from baseline. The TNSS is an instrument used to collect patient self-rated severity of rhinorrhea, nasal congestion, nasal itching and sneezing. In this study, a reflective score will be collected, in which the subject will be asked to evaluate symptom severity over the preceding 12 hours. Symptom severity is rated on a 4-point scale of 0 (absent symptoms), 1 (mild symptoms), 2 (moderate symptoms, or 3 (severe symptoms), with the total score therefore ranging from 0 to 12. A negative change reported for the change from baseline indicates an improved outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wolf, MD, Study Director — Aerin Medical, Inc.
Locations (5):
- United States (5):
  - Colorado ENT and Allergy, Colorado Springs, Colorado
  - Advanced ENT and Allergy, New Albany, Indiana
  - Piedmont ENT Associates, Winston-Salem, North Carolina
  - Fort Worth ENT, Fort Worth, Texas
  - ENT and Allergy Associates of Texas, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No